CLINICAL TRIAL: NCT03982966
Title: The Effect of the of Omega 3 Fatty Acids on the Vascular Calcification Biomarkers Fetuin A and Osteoprotegerin in Patients With Chronic Renal Failure Undergoing Hemodialysis.
Brief Title: Effect of Omega 3 Fatty Acids on the Vascular Calcification Biomarkers Fetuin A and Osteoprotegerin in Patients With CRF
Acronym: CRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Clinical Pharmacy Lecturer, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: omega 3 fatty acids on CRF
Record Dates: First submitted 2019-06-09; First posted 2019-06-12 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Intervention Model Description: enrolled patients will be divided into 2 groups, Group 1 will be 40 patients that will take omega 3fatty acids and Group 2 will be 20 patients served as control will not take omega 3 fatty acids.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 (Experimental): Group 1 will be 40 patients that will take Omega 3 fatty acids (fish oil)
  Interventions: Dietary Supplement: Omega 3 fatty acids (fish oil) 1000 mg/day oral
- Control (No Intervention): 20 patients will not take omega 3 fatty acids.

INTERVENTIONS:
Dietary Supplement: Omega 3 fatty acids (fish oil) 1000 mg/day oral — Omega 3 fatty acids (fish oil) 1000 mg/day oral
  Arms: Omega 3

SUMMARY:
study the effect of omega 3fatty acids on the vascular calcification biomarkers Fetuin -A and Osteoprotegerin (OPG) in dialysis patients.

DETAILED DESCRIPTION:
2-All Participants agreed to take part in this clinical research and provide informed consent.

3-Patients undergo both undergo hemodialysis (HD) will be enrolled from dialysis unit in al Moussa Hospital Alexandria.

4-Serum samples will be collected for measuring the biomarkers. 5-Our design is randomized, controlled, open-intervention study. 6- All enrolled patients will be divided into 2 groups, Group 1 will be 40 patients that will take omega 3fatty acids and Group 2 will be 20 patients will not take omega 3 fatty acids.

7-All patients will be followed up during 6 months' period. 8-Statsicial tests appropriate to the study design will be conducted to evaluate the significance of the results.

9-Measuring outcome: the primary outcome is the increase of the serum levels of the vascular calcification biomarkers after 6months.

10-Results, conclusions, discussion and recommendations will be given.

Inclusion criteria:

* 60 hemodialysis patients, (20-80) years old.
* Enrolled HD patients received regular HD 3 times weekly (on chronic maintenance for at least 6months).

Exclusion Criteria:

People with active infections (fever or any evidence of infections), known malignancy, connective tissue disorders, immunosuppressive therapy, and inflammatory diseases, current use of warfarin ,history of fish oil/omega 3 allergies were excluded.

Methodology:

* Feutin-A and Osteoprotegrin (OPG) will be determined by ELISA.
* Serum lipid levels, phosphorus, calcium, Parathormone (i-PTH), alkaline phosphatase, albumin and creatine levels.
* BMI

ELIGIBILITY:
Inclusion Criteria:

* 60 hemodialysis patients, (20-80) years old.
* Enrolled HD patients received regular HD 3 times weekly (on chronic maintenance for at least 6 months).

Exclusion Criteria:

* People with active infections (fever or any evidence of infections), known malignancy, connective tissue disorders, immunosuppressive therapy, and inflammatory diseases, current use of warfarin ,history of fish oil/omega 3 allergies were excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Feutin-A Level | six months
  vascular calcification biomarkers
Osteoprotegrin | six months
  vascular calcification biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Lecturer, Study Chair — Clinical Pharmacy Lecturer
Locations (1):
- al Mowassah Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] London GM, Marchais SJ, Guerin AP. Arterial stiffness and function in end-stage renal disease. Adv Chronic Kidney Dis. 2004 Apr;11(2):202-9. doi: 10.1053/j.arrt.2004.02.008. PMID 15216492
- [Background] Sigrist MK, Levin A, Er L, McIntyre CW. Elevated osteoprotegerin is associated with all-cause mortality in CKD stage 4 and 5 patients in addition to vascular calcification. Nephrol Dial Transplant. 2009 Oct;24(10):3157-62. doi: 10.1093/ndt/gfp253. Epub 2009 Jun 2. PMID 19491380